CLINICAL TRIAL: NCT06382779
Title: Proximal Humerus Reconstruction After Resection for Tumors : Comparison Between Allograft Prosthetic Composite and Cement Sleeve Prosthetic Composite
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, PEDUZZI Lisa, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI057
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Disease
Keywords: shoulder arthroplasty; reverse shoulder arthroplasty; allograft prosthetic composite

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- allograft prosthetic composite: patients treated with resection and reconstruction with reverse prostheses included in cryopreserved allografts
  Interventions: Procedure: reverse shoulder arthroplasty
- cement sleeve: patients treated with resection and reconstruction with suspended prostheses with proximal metaphyseal reconstruction using a cement sleeve
  Interventions: Procedure: reverse shoulder arthroplasty

INTERVENTIONS:
Procedure: reverse shoulder arthroplasty — resection of proximal humeral tumors and reconstruction with reverse shoulder arthroplasty

SUMMARY:
Proximal humerus is a common site for primary bone tumors and metastatic disease. Reconstruction with reverse shoulder arthroplasty (RSA) after resection is a surgical challenge and presented high risk of complication. The options for reconstruction after proximal humerus tumor resection are limited, and depend on the soft tissue conditions and bone loss. The most commonly used techniques include long cemented stem alone (in case of limited resection), allograft prosthetic composite (APC), massive prosthesis. In some cases two step procedure are performed : first step is resection and RSA with cement sleeve, and second step is APC or massive prosthesis.

DETAILED DESCRIPTION:
Theses surgical options are complex, technically challenging, and at risk of complications (dislocation, infections, allograft pseudarthrosis…). High complication rate, length of the surgical procedure and post-operative recovery are a concern for theses frail patients.

Timing before being able to schedule the intervention (selection of the appropriately sized allograft, restricted access to grafts…) is also an issue. Postponing cancer resection surgery increases the risk of both local and distant tumor invasion. In case of secondary bone tumors, surgery is often decided for pain relief rather than with a curative intent. In cases where rapid bone graft is not available, and urgent surgery is required for pain or for oncological reasons, the bone loss can be compensated for by a temporary cement sleeve . In some cases, either because life expectancy has improved or has been longer than anticipated, or because the patient declined a second surgery for the implantation of an allograft, some patients can stay with the reconstruction with a long-cemented stem and cement sleeve.

The objective of this study was to compare functional outcomes and complications between APC and cement sleeve reconstruction. Our hypothesis was that, in cases of proximal humerus resection for tumors, reverse prostheses included in cryopreserved allografts would yield better clinical results and greater longevity than suspended prostheses with proximal metaphyseal reconstruction using a cement sleeve.

ELIGIBILITY:
Inclusion Criteria:

* tumors of proximal humerus
* Malawer type I resection of this tumors
* primary reconstruction

Exclusion Criteria:

* resection and reconstruction by prosthesis alone
* resection and hemiarthroplasty reconstruction
* resection and revision protheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for tumors of proximal humerus, who underwent a Malawer type I resection of this tumors
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Constant score | through clinical completion an average of 2 years
  Shoulder functional evaluation score : between 6 points ( worse outcome) and 100 points (better outcome)

SECONDARY OUTCOMES:
complication | through clinical completion an average of 5 years
  dislocation, infection,
mortality | through clinical completion an average of 5 years
  death: intervention-related or non-intervention-related, cause of death, delay of death
revision | through clinical completion an average of 5 years
  reoperation (with or without implant extraction), cause of revision, delay of revision

CONTACTS AND LOCATIONS:
Overall Officials: Francois SIRVEAUX, Study Chair — Central Hospital, Nancy, France
Locations (1):
- CHRU - Centre chirurgical emile galle, Nancy, France